CLINICAL TRIAL: NCT02201758
Title: Flaxseed Lignan-enriched Complex (FLC) for the Treatment of Patients With Mild to Moderately Severe Ulcerative Colitis (UC): A Pilot Assessment.
Brief Title: Flaxseed Lignan-Enriched Complex (FLC) for the Treatment of Patients With Ulcerative Colitis (UC): A Pilot Assessment
Acronym: FLC&UC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researchers decided to withdrawn the study due unavialble FLC
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Sharyle Fowler, M.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio 14-128
Record Dates: First submitted 2014-07-18; First posted 2014-07-28 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease (IBD); ulcerative colitis (UC); flaxseed lignan-enriched complex (FLC)
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Flaxseed Lignan-Enriched Complex (FLC) vs. placebo
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will consist of unflavored whey protein (manufactured by Natural Factors®)
  Interventions: Other: Placebo
- flaxseed lignan-enriched complex (FLC) (Experimental): Subjects will undergo treatment with FLC for an 8-week period; participants will take 300 mg flaxseed lignan-enriched complex (FLC) taken orally twice daily
  Interventions: Dietary Supplement: Flaxseed lignan-enriched complex (FLC)

INTERVENTIONS:
Dietary Supplement: Flaxseed lignan-enriched complex (FLC) — Subjects will undergo treatment with FLC for an 8-week period; participants will take 300 mg flaxseed lignan-enriched complex (FLC) taken orally twice daily
  Arms: flaxseed lignan-enriched complex (FLC)
Other: Placebo — Placebo will consist of unflavored whey protein (manufactured by Natural Factors®)
  Other Names: Placebo Comparator: Placebo
  Arms: Placebo

SUMMARY:
This study proposes to examine the effect of diet as a modifiable risk factor among patients with ulcerative colitis (UC). Flax seeds contain many bioactive constituents which have anti-oxidative, anti-inflammatory, and anti-carcinogenic effects. These bioactive compounds represent novel classes of pharmacologically active compounds which may represent new options to treat chronic disease of the gastrointestinal tract. Participants with mild to moderately severe UC will supplement their current medications with flaxseed lignan-enriched complex (FLC). This is a 12 week double blind placebo controlled study with assessment throughout. Stool and blood samples (biomarkers) as well as bowel assessment via sigmoidoscopy will be evaluated before and after the intervention. The treatment arm consists of 300 mg FLC taken orally twice daily.

DETAILED DESCRIPTION:
This project is a single centre, randomized, placebo-controlled pilot study in which subjects recruited to the study will undergo treatment with FLC for an 8-week period. The investigators will recruit patients with mild to moderately severe, left-sided or pan-colonic UC (Mayo Score 3 - 10 points). All participants will have vitamin D status evaluated at baseline and clinically indicated laboratory investigations including complete blood count (CBC), liver enzymes and serologic inflammatory marker high sensitivity c-reactive protein (hsCRP). Participants will be evaluated at weeks 0, 2, 4 and 8 during the treatment period and at week 10 at follow-up. Exclusion criteria will include a colectomy, positive stool culture for common bacterial pathogens, a history of drug or alcohol abuse, mental illness, concomitant immunological, hematologic or neoplastic disease, hepatic insufficiency, cardiac insufficiency, pregnancy, treatment with anti-tumor necrosis factor agents within 3 months, local steroids in the preceding 30 days, and antibiotics less than 15 days before screening. Participants may continue concomitant medications at stable dosages for at least 12 weeks before screening (medications include mesalamine, thiopurines, methotrexate, and probiotics). Participants will continue current medication if she/he is stable with it; no washout period is required. FLC will be a supplement therapy; dosages of concomitant medications must be maintained constant throughout the study.

The introduction of biologics, steroids, or antibiotics or any dose increase of existing medication during the study will be considered a treatment failure. Subjects meeting inclusion and exclusion criteria will be randomized by a computer-generated algorithm in a 1:1 fashion to one of two treatment arms. Treatment Arm 1 will consist of 300 mg FLC taken orally twice daily. The 600 mg dose of FLC is based on clinical research that suggests a minimum dose of 500 mg/day dose of FLC is tolerable and necessary to observe significant health benefits (i.e. reduction of cardiovascular risk). The placebo will consist of unflavored whey protein (manufactured by Natural Factors®). FLC and placebo packets will be prepared by study personnel in the College of Pharmacy and Nutrition under the supervision of a licensed pharmacist. Participants and investigators will be blinded to treatment allocation.

The primary outcome of interest will be the comparative proportion of subjects who complete the study at week 8. Secondary endpoints will include the proportion of week 8 clinical responders (as defined by a Mayo Score reduction of ≥ 3 points) and the proportion of subjects with a post-therapy fecal calprotectin (Cp) concentration ≤ 150 μg/g at week 8.

The study will be powered to detect the primary endpoint, which is the proportion of subjects completing the study at week 8 in the FLC versus the placebo-treated group. Power calculations based upon a two-sided 95% confidence interval (α = 0.05) with an estimated study completion rate of 0.40 in the placebo-treated group and 0.80 in the FLC treated group indicate that 28 subjects will need to be recruited per group in order to detect a difference (β = 0.80). Relevant covariates including smoking status, gender, age, disease duration and disease severity will be compared between intervention and placebo groups using the χ2 test of independence for categorical variables and ANOVA for continuous variables. Missing data will be handled through multiple imputation techniques with appropriate sensitivity analysis to investigate the effects of different imputation methods.

The use of the FLC complex holds promise in attenuating inflammation found in IBD. The investigators suspect that using FLC in patients with mild to moderately severe UC will be well-tolerated and efficacious. Data derived from this pilot study will inform planned future national, double-blind, placebo-controlled intervention trials on the therapeutic potential of flaxseed derived products in IBD and will be the first study of its kind to investigate FLC as therapy in IBD.

The data derived from this pilot study will help to determine whether flaxseed derived bioactive is a safe and cost-effective alternative therapeutic option for the treatment of patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years and above
2. Patients diagnosed with mild to moderately severe, left-sided or pan-colonic UC (Mayo Score 3 - 10 points)
3. Baseline vitamin D status and clinically indicated laboratory investigations such as CBC, liver enzymes and serologic inflammatory marker high sensitivity c-reactive protein (hsCRP).

Exclusion Criteria:

Patients with the following conditions will be excluded:

* colectomy
* positive stool culture for common bacterial pathogens
* history of drug or alcohol abuse
* mental illness
* concomitant immunological
* hematologic or neoplastic disease
* hepatic insufficiency
* cardiac insufficiency
* pregnancy
* treatment with anti-tumor necrosis factor agents within 3 months
* local steroids in the preceding 30 days and antibiotics less than 15 days before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete study period | 8 weeks
  The primary outcome of interest will be the comparative proportion of subjects who complete the study at week 8.

SECONDARY OUTCOMES:
Proportion of clinical responders | 8 weeks
  Proportion of week 8 clinical responders is defined by a Mayo Score reduction of ≥ 3 points

OTHER OUTCOMES:
Post-therapy fecal calprotectin (Cp) | 8 weeks
  Proportion of subjects with a post-therapy fecal calprotectin (Cp) concentration equal or less than 150 mg/g at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Sharyle Fowler, MD,FRCPS, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada